CLINICAL TRIAL: NCT00195052
Title: Intraoperative Optical Mapping of Human Epileptiform and Functional Cortex
Brief Title: Intrinsic Optical Imaging Study to Map Neocortical Seizure in Human Epilepsy Patients
Status: Terminated | Type: Observational
Why Stopped: The study is terminating prematurely as Dr. Schwartz is no longer at WCM, and the study cannot feasibly be completed in his absence.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0102004808
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
Keywords: epilepsy; optical imaging; optical mapping
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epilepsy Patients
  Interventions: Diagnostic Test: Intrinsic signal imaging of human cortex

INTERVENTIONS:
Diagnostic Test: Intrinsic signal imaging of human cortex — Light is shined on the brain at 540 nm and 610 nm and images are acquired at 10 frames per second.

SUMMARY:
The purpose of this study is to develop a technique for the intraoperative identification of human functional and epileptiform cortex using intrinsic signal imaging. The investigators propose that the ability to optically monitor neuronal activity in a large area of cortex in "real-time" will be a more sensitive and time-saving method than the electrical methods currently available. The applications of this technique will not only theoretically increase the safety and efficacy of many of neurosurgical procedures, but will be useful as an investigational tool to study human cortical physiology.

DETAILED DESCRIPTION:
Epilepsy is a disease affecting 1-2% of the population. Currently, the only known cure for epilepsy is surgery, which is much more effective at eliminating seizures arising from the medial temporal lobe compared with the neocortex. The problem with neocortical epilepsy is that the population of neurons underlying each epileptiform discharge varies over time. In addition, the spatial relationship between interictal events and the ictal onset zones, which are critical in defining the region of epileptogenesis, is not well understood and essential to the surgical treatment of epilepsy. Electrophysiological recording methods, although currently the "gold standard" in mapping epilepsy, are inadequate to address these questions based on restrictions due to volume conduction or sampling limitations. Optical recording techniques can overcome many of these limitations by sampling large areas of cortex simultaneously to provide information about blood flow, metabolism and extracellular fluid shifts that are intimately related to excitatory and inhibitory neuronal activity. In fact, optical recordings may actually be more sensitive to certain aspects of epileptic activity than electrophysiologic recordings. The goal will be to translate these findings into the operating room and map human neocortical epilepsy with the same optical techniques. Outcome following surgical resections to treat neocortical epilepsy will be correlated with the optical maps to determine the utility of intrinsic signal imaging in guiding brain surgery. These experiments will set the groundwork for implementing optical recordings in general clinical practice as a novel technique for mapping and predicting human seizures.

ELIGIBILITY:
Inclusion Criteria:

* Medically intractable epilepsy
* Subjects undergoing neurosurgical operations requiring cortical mapping

Exclusion Criteria:

* Subjects NOT undergoing neurosurgical operations requiring cortical mapping.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient, who is going to undergo a neurosurigcal procedure which will require intraoperative brain mapping to determine the brain organization, is the potential study subject.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2025-04 (Actual); Study Completion 2025-04 (Actual)

PRIMARY OUTCOMES:
Positive identification of language areas with optical imaging | During surgery (20-30 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore H Schwartz, MD, Principal Investigator — Weill Cornell Medical College/New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No